CLINICAL TRIAL: NCT04590898
Title: Safety and Feasibility of Peri-device Leakage Closure After Left Atrial Appendage Occlusion
Brief Title: Peri-device Leakage Closure After LAAO
Status: Completed | Type: Observational
Sponsor: Cardiovascular Center Frankfurt (Other)
Responsible Party: Sponsor
Other Study IDs: CVC-002
Record Dates: First submitted 2020-10-01; First posted 2020-10-19 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Atrial Fibrillation; Stroke; Bleeding; Leakage of Cardiac Device
Keywords: left atrial appendage occlusion; peri-device leakage; stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- significant peri-device leakage after LAA occlusion: Peri-device leakage closure after left atrial appendage occlusion
  Interventions: Device: Peri-device leakage closure after left atrial appendage occlusion

INTERVENTIONS:
Device: Peri-device leakage closure after left atrial appendage occlusion — Peri-device leakage closure after left atrial appendage occlusion

SUMMARY:
The investigators thought to evaluate the safety and feasibility of peri-device leakage closure after left atrial appendage occlusion (LAAO, either surgical or interventional) with different devices.

DETAILED DESCRIPTION:
The global burden of atrial fibrillation (AF) is high and thromboembolic stroke may be one of the fatal complications. Oral anticoagulation has been the mainstay therapy for decades to mitigate stroke risk. However, in poor candidates for long-term anticoagulation non-pharmacological stroke prevention with percutaneous left atrial appendage occlusion (LAAO) is a considerable treatment option. LAA shape and size varies widely and incomplete LAA closure or new leaks, due to LAA remodeling after the procedure, are observed in up to 30% of patients. Those leaks may cause turbulent flow and increase the risk for thrombus formation and subsequent thromboembolic events. However, the clinical significance after percutaneous LAAO has yet to be determined.

If significant leaks are present, patients usually remain on oral anticoagulation. In very few cases, an interventional approach is used to close peri-device leaks.

This is the first systematic study, trying to include a respectable number of patients who underwent peri-device leakage closure after LAAO. In this multi-center, collaborative study the investigators aim to identify different peri-device leak closure strategies with associated clinical outcomes and evaluate safety and feasibility of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients after interventional or surgical left atrial appendage occlusion with severe leakage, who underwent interventional peri-device leakage closure

Exclusion Criteria:

* n/a

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after interventional or surgical left atrial appendage occlusion with severe leakage, who underwent interventional peri-device leakage closure
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2020-09-27 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Procedural mortality | In-hospital stay, assessed up to 30days
  Rate of all-cause mortality during the index procedure, number of participants experiencing a procedure-related death within 30days or during in-hospital stay for the index procedure (if>30days)
Procedure-related clinically relevant pericardial effusion | In-hospital stay, assessed up to 30days
  Number of participants experiencing pericardial effusion with hemodynamic relevance, treated with therapeutic pericardiocentesis or surgical intervention, requiring blood transfusion or resulting in shock and/or death, which was procedure related
Procedure-related ischemic stroke | In-hospital stay, assessed up to 30days
  Number of participants experiencing an acute episode of focal cerebral, spinal, or retinal dysfunction caused by infarction of central nervous system tissue, which was procedure related

SECONDARY OUTCOMES:
Bleeding complications | through study completion, an average of 1 year
  Number of participants experiencing bleeding complications evaluated by using VARC-2 criteria with LAAO specific modifications (after the Munich consensus document on definitions, endpoints, and data collection requirements for clinical studies)
Vascular access site complications | during procedure, assessed up to 7 days
  Number of participants experiencing retroperitoneal haematoma, AV-fistula, arterial complications, venous complications, symptomatic peripheral ischemia, nerve injury with clinical symptoms >24h, vascular surgical repair at access site, pulmonary embolism, ipsilateral deep vein thrombosis, access site-related infection requiring iv. antibiotics or extended hospitalization
Liver- and kidney failure associated with the procedure | In-hospital stay, assessed up to 30days
  Number of participants experiencing liver- and kidney failure potentially associated with the procedure evaluated by using the definitions of Munich consensus document on definitions, endpoints, and data collection requirements for clinical studies
Device-associated complications | through study completion, an average of 1 year
  Number of participants experiencingdevice migration, perforation, laceration, erosion, device infection, pericarditis, device-related thrombus and persistent or occurrence of new peri-device leakage
Ischemic stroke or transitory ischemic attack | through study completion, an average of 1 year
  Number of participants experiencing an acute episode of focal cerebral, spinal, or retinal dysfunction caused by infarction of central nervous system tissue not directly related to the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Piayda, Study Chair — University Hospital Düsseldorf and Cardio Vascular Center Frankfurt
Locations (16):
- United States (7):
  - • Banner University Medical Center Phoenix, Phoenix, Arizona
  - Scripps Health, La Jolla, California
  - Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - Mayo Clinic Hospital - Saint Mary's Campus, Rochester, Minnesota
  - Vanderbilt Heart Institute, Nashville, Tennessee
  - Austin Heart, Austin, Texas
  - University of Utah Hospital, Salt Lake City, Utah
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet Copenhagen, Copenhagen
- Germany (3):
  - Cardio Vascular Center Frankfurt, Frankfurt am Main, Hesse
  - Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Universitätsmedizin Berlin - Campus Benjamin Franklin (CBF), Berlin
- Poznan University of Medical Sciences, Poznan, Poland
- Hospital Universitario de Salamanca, Salamanca, Spain
- Inselspital Bern, Bern, Switzerland
- Nuffield Health, Headington, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided